CLINICAL TRIAL: NCT01302912
Title: Lymphoma in the Orbit
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: USZ-OALs-Register
Record Dates: First submitted 2011-02-23; First posted 2011-02-24 (Estimated); Last update posted 2011-11-04 (Estimated); Status verified 2011-11

CONDITIONS: Ocular Adnexal Mucosa-Associated Lymphoid Tissue Lymphoma
Keywords: ocular adnexal lymphomas

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

INTERVENTIONS:
Procedure: Lymphoma-Biopsy — Patients after biopsy of orbital lymphoma

SUMMARY:
Imaging techniques have considerably improved over the last decades and ocular adnexal lymphomas (OALs) nowadays can be detected. As major advances in immunophenotyping and molecular diagnostics in histology have been achieved offering an accurate diagnosis, the investigators would like to introduce that surgical biopsy of an orbital lymphoma becomes crucial for the possibility of a correct diagnosis and proper treatment. As radiotherapy accomplished great preciseness as well and OALs respond excellently to radiation, this therapy should be the treatment of choice in local defined lymphomas instead of blind treatment with steroids. Radiation results in great local control rates of 85% to 100%

* Trial with surgical intervention

ELIGIBILITY:
Inclusion criteria: - both genders

* >17 years of age
* underwent biopsy of an ocular adnexal lymphoma between 01/2006 and 12/2010 at the University Hospital Zurich, Division of Ophthalmology
* diagnosis histologically proven

Exclusion criteria:

* less than 18 years of age
* patient underwent no MRI before surgery (biopsy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient, who underwent biopsy of an ocular adnexal lymphoma between 01/2006 and 12/2010 at the University Hospital Zurich, Division of Ophthalmology
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2011-02; Study Completion 2012-05 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Karla Chaloupka, MD, Principal Investigator — University Hospital Zurich, Ophtalmic Clinic
Locations (1):
- University Hospital Zurich, Ophthalmic Clinic, Zurich, Canton of Zurich, Switzerland